CLINICAL TRIAL: NCT01547741
Title: A Phase III Clinical Trial Comparing the Combination of Docetaxel Plus Cyclophosphamide to Anthracycline-Based Chemotherapy Regimens for Women With Node-Positive or High-Risk Node-Negative, HER2-Negative Breast Cancer
Brief Title: Docetaxel and Cyclophosphamide Compared to Anthracycline-Based Chemotherapy in Treating Women With HER2-Negative Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP-B-49; NCI-2012-00701 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; HER2-negative breast cancer; progesterone receptor-negative breast cancer; progesterone receptor-positive breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Docetaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Anthracycline-based chemotherapy (Active Comparator): 4 anthracycline-based chemotherapy regimens (Regimens A, B, C, or D).
  Regimen A (TAC): 75 mg/m2 docetaxel (T) + 50 mg/m2 doxorubicin (A) + 500 mg/m2 cyclophosphamide (C) IV every 3 weeks for 6 cycles.
  Regimen B (AC then WP): 60 mg/m2 doxorubicin (A) + 600 mg/m2 cyclophosphamide (C) every 3 weeks for 4 cycles followed by weekly paclitaxel (WP) 80 mg/m2 IV every week for 12 doses.
  Regimen C (DD AC then WP): 60 mg/m2 doxorubicin + 600 mg/m2 cyclophosphamide every 2 weeks for 4 cycles followed by weekly paclitaxel 80 mg/m2 IV every week for 12 doses.
  Regimen D (DD AC then DD P): 60 mg/m2 doxorubicin + 600 mg/m2 cyclophosphamide every 2 weeks for 4 cycles followed by paclitaxel (P) 175 mg/m2 IV every 2 weeks for 4 cycles.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Paclitaxel
- Arm 2: docetaxel + cyclophosphamide (Active Comparator): TC: 75 mg/m2 docetaxel and 600 mg/m2 cyclophosphamide IV every 3 weeks for 6 cycles
  Interventions: Drug: Cyclophosphamide; Drug: Docetaxel

INTERVENTIONS:
Drug: Doxorubicin
  Other Names: adriamycin
  Arms: Arm 1: Anthracycline-based chemotherapy
Drug: Cyclophosphamide
Drug: Docetaxel
Drug: Paclitaxel
  Arms: Arm 1: Anthracycline-based chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of breast cancer cells, either by killing the cells or by stopping them from dividing. Giving the drugs in different combinations may kill more breast cancer cells. Giving combination chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This randomized phase III trial is studying different combination chemotherapy regimens and their side effects and comparing how well they work in treating women with non-metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if the docetaxel and cyclophosphamide (TC) regimen is non-inferior to the anthracycline-based chemotherapy regimens in terms of invasive disease-free survival (DFS) by combining B-49 data with the docetaxel, doxorubicin, and cyclophosphamide (TAC) and TC arms of NSABP B-46-I/US Oncology Research, Inc.(USOR) 07132 and the data from USOR 06-090.

Secondary

* To determine rates of DFS-ductal carcinoma in situ (DCIS) for the TC and anthracycline-based chemotherapy regimens.
* To determine rates of overall survival (OS) for the TC and anthracycline-based chemotherapy regimens.
* To determine rates of recurrence-free interval (RFI) for the TC and anthracycline-based chemotherapy regimens.
* To evaluate the toxicity associated with each of the regimens.
* To determine the role of TOP2A in prognosis and prediction of degree of benefit from anthracycline-based chemotherapy over TC. (exploratory)
* To develop predictive markers for benefit from doxorubicin. (exploratory)

OUTLINE: This is a multicenter randomized study. Patients are stratified according to number of positive nodes (0 vs 1-3 vs 4-9 vs 10+) and hormone-receptor status (estrogen receptor [ER] and/or progesterone receptor [PgR] positive vs ER and PgR negative). Patients are randomized to 1 of 2 treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The tumor must be unilateral invasive adenocarcinoma of the breast on histologic examination.
* The breast cancer must be Human Epidermal Growth Factor Receptor 2 (HER2)-negative based on current American Society of Clinical Oncology (ASCO)/CAP Guideline Recommendations for Human Epidermal Growth Factor Receptor 2 Testing in Breast Cancer. If the result of the in situ hybridization testing (FISH, chromagen in situ hybridization [CISH], or other) is equivocal, the patient is eligible if there is no plan to administer HER2-targeted therapy.
* All of the following staging criteria must be met according to American Joint Committee on Cancer (AJCC) criteria:

  * By pathologic evaluation, primary tumor must be pT1-3;
  * By pathologic evaluation, ipsilateral nodes must be pN0, pN1 (pN1mi, pN1a, pN1b, pN1c), pN2a, pN3a, or pN3b.
  * If pN0, at least one of the following criteria must be met:
  * ER negative and PgR negative; or
  * Pathologic tumor size greater than 2.0 cm; or
  * T1c (pathologic tumor size greater than 1.0 cm but less than or equal to 2.0 cm) and ER positive (PgR status may be positive or negative) and either grade 3 histology or Oncotype DX® Recurrence Score of greater than or equal to 25.
* Patients must have undergone either a total mastectomy or breast-conserving surgery (lumpectomy).
* For patients who undergo lumpectomy, the margins of the resected specimen must be histologically free of invasive tumor and ductal carcinoma in situ (DCIS) as determined by the local pathologist. If pathologic examination demonstrates tumor at the line of resection, additional operative procedures must be performed to obtain clear margins. If tumor is still present at the resected margin after re-excision(s), the patient must undergo total mastectomy to be eligible. (Patients with margins positive for lobular carcinoma in situ [LCIS] are eligible without additional resection.)
* For patients who undergo mastectomy, margins must be histologically free of invasive tumor and DCIS.
* Patients must have completed one of the following procedures for evaluation of pathologic nodal status:

  * Sentinel lymphadenectomy alone if pathologic nodal staging based on sentinel lymphadenectomy is pN0, pN1mi, or pN1b;
  * Sentinel lymphadenectomy alone if pathologic nodal staging based on sentinel lymphadenectomy is pN1a limited to 1 or 2 positive nodes and primary tumor is T1 or T2 by pathologic evaluation;
  * Sentinel lymphadenectomy followed by removal of additional non-sentinel lymph nodes if the sentinel node (SN) is positive; or
  * Axillary lymphadenectomy with or without SN isolation procedure.
* The interval between the last surgery for breast cancer (treatment or staging) and randomization must be no more than 84 days.
* Patients must have ER analysis performed on the primary tumor prior to randomization. Breast cancer must be assessed for ER status by current ASCO/CAP Guideline Recommendations for hormone receptor testing. If negative for ER, assessment of PgR must also be performed according to current ASCO/CAP Guideline Recommendations for hormone receptor testing. (Either a core biopsy or surgical resection specimen can be used for ER/PgR testing.)
* The most recent postoperative blood counts, performed within 6 weeks prior to randomization, must meet the following criteria:

  * absolute neutrophil count (ANC) must be greater than or equal to 1200/mm3;
  * platelet count must be greater than or equal to 100,000/mm3; and
  * hemoglobin must be greater than or equal to 10 g/dL.
* The following criteria for evidence of adequate hepatic function must be met based on the results of the most recent postoperative tests performed within 6 weeks prior to randomization:

  * total bilirubin must be less than or equal to upper limit of normal (ULN) for the lab unless the patient has a bilirubin elevation greater than ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and
  * alkaline phosphatase must be less than or equal to 2.5 x ULN for the lab; and
  * aspartate transaminase (AST) must be less than or equal to 1.5 x ULN for the lab.
  * Alkaline phosphatase and AST may not both be greater than the ULN. For example, if the alkaline phosphatase is greater than the ULN but less than or equal to 2.5 x ULN, then the AST must be less than or equal to the ULN. If the AST is greater than the ULN but less than or equal to 1.5 x ULN, then the alkaline phosphatase must be less than or equal to ULN.
  * Note: If alanine aminotransferase (ALT) is performed instead of AST (per institution's standard practice), the ALT value must be less than or equal to 1.5 x ULN; if both were performed, the AST must be less than or equal to 1.5 x ULN.
* Patients with AST or alkaline phosphatase greater than ULN are eligible for inclusion in the study if liver imaging (CT, MRI, PET-CT, or PET scan performed within 90 days prior to randomization) does not demonstrate metastatic disease and the requirements for adequate hepatic function as described above are met.
* Patients with alkaline phosphatase that is greater than ULN but less than or equal to 2.5 x ULN are eligible for inclusion in the study if a bone scan, PET-CT scan, or PET scan performed within 90 days prior to randomization does not demonstrate metastatic disease.
* The most recent postoperative serum creatinine performed within 6 weeks prior to randomization must be less than or equal to ULN for the lab.
* Left ventricular ejection fraction (LVEF) assessment by 2-D echocardiogram or multigated acquisition (MUGA) scan must be performed within 90 days prior to randomization. The LVEF must be greater than or equal to 50% regardless of the facility's lower limit of normal (LLN). (If the facility performing the assessment has not reported the LVEF as a whole number, decimals reported as greater than or equal to 5 should be rounded up and decimals reported as less than 5 should be rounded down.)

Exclusion criteria:

Patients with one or more of the following conditions are ineligible for this study.

* T4 tumors including inflammatory breast cancer.
* Definitive clinical or radiologic evidence of metastatic disease. (Chest imaging [mandatory for all patients] and other imaging [if required] must have been performed within 90 days prior to randomization.)
* Synchronous or previous contralateral invasive breast cancer. (Patients with synchronous and/or previous contralateral DCIS are eligible.)
* Any history of ipsilateral invasive breast cancer or ipsilateral DCIS.
* History of non-breast malignancies within 5 years prior to randomization, except for the following: carcinoma in situ of the cervix, colorectal carcinoma in situ, melanoma in situ, and basal cell and squamous cell carcinomas of the skin.
* Previous therapy with anthracyclines or taxanes for any malignancy.
* Chemotherapy administered for the currently diagnosed breast cancer prior to randomization.
* Continued endocrine therapy such as raloxifene or tamoxifen (or other SERM) or an aromatase inhibitor. Patients are eligible if these medications are discontinued prior to randomization.
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormone replacement therapy. Patients are eligible if these medications are discontinued prior to randomization.
* Known active hepatitis B or hepatitis C with abnormal liver function tests.
* Cardiac disease (history of and/or active disease) that would preclude the use of the drugs included in the treatment regimens. This includes but is not confined to:

  * Active cardiac disease
  * angina pectoris that requires the use of anti-anginal medication;
  * ventricular arrhythmias except for benign premature ventricular contractions;
  * supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication;
  * conduction abnormality requiring a pacemaker;
  * valvular disease with documented compromise in cardiac function;
  * symptomatic pericarditis.
  * History of cardiac disease
  * myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular function;
  * history of documented congestive heart failure (CHF);
  * documented cardiomyopathy.
* Whole breast radiation therapy (RT) prior to randomization or partial breast RT that cannot be completed on or before the date of randomization.
* Intrinsic lung disease resulting in dyspnea.
* Unstable diabetes mellitus.
* Active infection or chronic infection requiring suppressive antibiotics.
* History of a major organ allograft or condition requiring chronic immunosuppression, e.g., kidney, liver, lung, heart, bone marrow transplant, or autoimmune diseases. (Patients who have received corneal transplants, cadaver skin, or bone transplants are eligible.)
* Nervous system disorder (paresthesia, peripheral motor neuropathy, or peripheral sensory neuropathy) greater than or equal to grade 2, per the NCI CTCAE v4.0.
* Conditions that would prohibit administration of corticosteroids.
* Chronic daily treatment with corticosteroids (dose of greater than or equal to 10 mg/day methylprednisolone equivalent) (excluding inhaled steroids).
* History of hypersensitivity reaction to drugs formulated with polysorbate 80.
* Pregnancy or lactation at the time of study entry. (Note: Pregnancy testing must be performed within 2 weeks prior to randomization according to institutional standards for women of childbearing potential.)
* Other non-malignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
* Use of any investigational product within 30 days prior to randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1871 (Actual)
Dates: Start 2012-04; Primary Completion 2022-05 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (IDFS) | Assessed before each cycle of chemotherapy, 3-4 weeks after completion of chemotherapy, every 6 months through 5 years and yearly years 6-10.
  The time to local recurrence following mastectomy, invasive local recurrence in the ipsilateral breast following lumpectomy, regional recurrence, distant recurrence, invasive contralateral breast cancer, second primary cancer (other than squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, colorectal carcinoma in situ, or lobular carcinoma in situ of the breast), or death from any cause prior to recurrence or second primary cancer.

SECONDARY OUTCOMES:
Disease-free survival (DFS-DCIS) | Assessed before each cycle of chemotherapy, 3-4 weeks after completion of chemotherapy, every 6 months through 5 years and yearly years 6-10.
  The time to local recurrence following mastectomy, local recurrence in the ipsilateral breast following lumpectomy (invasive or non-invasive), regional recurrence, distant recurrence, contralateral breast cancer (invasive or non-invasive), second primary cancer (other than squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, colorectal carcinoma in situ, or lobular carcinoma in situ of the breast), or death from any cause prior to recurrence or second primary cancer.
Overall survival (OS) | Assessed before each cycle of chemotherapy, 3-4 weeks after completion of chemotherapy, every 6 months through 5 years and yearly years 6-10.
  Time from randomization until death from any cause.
Recurrence-free interval (RFI) | Assessed before each cycle of chemotherapy, 3-4 weeks after completion of chemotherapy, every 6 months through 5 years and yearly years 6-10.
  Time from randomization until local, regional, or distant recurrence.
Toxicity of each regimen | Assessed before each cycle of chemotherapy, 3-4 weeks after completion of chemotherapy, every 6 months through 5 years and yearly years 6-10.
  Frequencies of adverse events categorized using the NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Molecular predictors of efficacy | Tissue sample collected at time of surgery
  To develop predictive markers for benefit from doxorubicin.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (915):
- United States (914):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arizona Oncology Associates-Biltmore Cancer Center, Phoenix, Arizona
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Sedona Medical Center, Sedona, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - NEA Baptist Clinic-Matthews, Jonesboro, Arkansas
  - Kaiser Anaheim Medical Center, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente Medical Group - Baldwin Park, Baldwin Park, California
  - Kaiser Foundation Hospital, Bellflower, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Epic Care-Dublin, Dublin, California
  - Northbay Cancer Center, Fairfield, California
  - Kaiser Permanente Hospital, Fontana, California
  - Kaiser Permanente, Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - California Cancer Center - North Fresno, Fresno, California
  - Kaiser Permanente, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente, Hayward, Hayward, California
  - Southern California Permanente Medical Group, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente, Los Angeles, California
  - Kaiser Permanente-West Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons Inc, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Epic Care-Oakland, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Feather River Cancer Center, Paradise, California
  - East Bay Medical Oncology Hematology Medical Associates Inc-Pleasant Hill, Pleasant Hill, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente Medical Center, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente at San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Kaiser Permanente Health Care, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente, Woodland Hills, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Saint Anthony Central Hospital, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - Bayhealth Medical Center at Kent General, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Saint Vincent's Medical Center, Jacksonville, Florida
  - Edna Williams Cancer Center at the Baptist Cancer Institute, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - The Watson Clinic, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Advanced Medical Specialties -North, Miami, Florida
  - Mount Sinai Medical Center CCOP, Miami Beach, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - M D Anderson Cancer Center- Orlando, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Sacred Heart Medical Oncology Group - Davis Highway, Pensacola, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Augusta Oncology Associates PC-Saint Sebastian, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Joseph's-Candler Health System, Savannah, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii Inc - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Idaho Urologic Institute PA, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Evanston CCOP-NorthShore University HealthSystem, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - FHN Leonard C. Ferguson Cancer Center, Freeport, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Medical and Surgical Specialists, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Adventist La Grange Memorial Hospital, La Grange, Illinois
  - North Shore Hematology Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Medical Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Hematology Oncology Consultants Limited, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Mid-Illinois Hematology Oncology Associates, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Cancer Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Foundation - Carle Cancer Center, Urbana, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc - State Boulevard, Fort Wayne, Indiana
  - Central Indiana Cancer Centers - Indianapolis, Indianapolis, Indiana
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Indiana University Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett, Lafayette, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Saint Anthony Memorial Health Center, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology-PC Westville, Westville, Indiana
  - McFarland Clinic, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Hematology Oncology Associates-Quad Cities, Bettendorf, Iowa
  - Helen G Nassif Community Cancer Center, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Promise Regional Medical Center-Hutchinson, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas City Cancer Center-West, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center-Shawnee Mission, Shawnee Mission, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Regional Medical Center, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Norton Health Care Pavilion - Downtown, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Clinic Foundation-Baton Rouge, Baton Rouge, Louisiana
  - Ochsner North Shore Medical Center, Covington, Louisiana
  - Interim LSU Public Hospital, New Orleans, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Clinic CCOP, New Orleans, Louisiana
  - Christus Schumpert Saint Mary's Place, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Mercy Hospital, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Maine Center for Cancer Medicine and Blood Disorders-Scarborough, Scarborough, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - The Union Memorial Hospital, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Maryland Oncology Hematology PA-Columbia, Columbia, Maryland
  - The Memorial Hospital at Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Berkshire Hematology Oncology PC, Pittsfield, Massachusetts
  - Jordan Hospital, Plymouth, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Great Lakes Cancer Institute, Clarkston, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Michigan State University - Breslin Cancer Center, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Great Lakes Cancer Institute-Lapeer Campus, Lapeer, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Mount Clemens Regional Medical Center, Mount Clemens, Michigan
  - Mercy Health Partners-Mercy Campus, Muskegon, Michigan
  - Memorial Healthcare Center, Owosso, Michigan
  - Northern Michigan Regional Hospital, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Mayo Clinic Health System in Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Forest General Hospital, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Saint John's Regional Medical Center, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Cancer Center - South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Clinic, Liberty, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Ozark Health Ventures LLC dba Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - Saint John's Hospital, Springfield, Missouri
  - Cox Medical Center, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Good Samaritan Hospital, Kearney, Nebraska
  - Lincoln Medical Education Foundation Cancer Resource Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium CCOP, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology PA, Concord, New Hampshire
  - New Hampshire Oncology Hematology Associates, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Cancer Institute of New Jersey At Hamilton, Hamilton, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - South Jersey Healthcare, Vineland, New Jersey
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC -Albany Medical Center, Albany, New York
  - New York Oncology Hematology PC - Amsterdam, Amsterdam, New York
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York PC, East Syracuse, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - Broome Oncology LLC, Johnson City, New York
  - Monter Cancer Center, Lake Success, New York
  - New York Oncology Hematology PC - Latham, Latham, New York
  - North Shore University Hospital, Manhasset, New York
  - North Shore-LIJ Health System CCOP, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Saint Francis, Poughkeepsie, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Alamance Regional Medical Center, Burlington, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Carolinas Medical Center - Northeast, Concord, North Carolina
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Carolinas Medical Center-Union, Monroe, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Cleveland Regional Medical Center, Shelby, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L Shepard Cancer Center, Washington, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Forsyth Memorial Hospital, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Akron City Hospital, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Health Partners Regional Medical Center, Elyria, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Mansfield General Hospital-MedCentral Health System, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Cancer Center-Strongsville, Strongsville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Cancer Center at Saint Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Specialty Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates-Mercy, Oklahoma City, Oklahoma
  - Natalie W Bryant Cancer Center, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Asante Health System, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Columbia River Oncology Program, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Mid-Columbia Medical Center, The Dalles, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - The Regional Cancer Center, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - PinnacleHealth Fox Chase Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Riddle Hospital, Media, Pennsylvania
  - Forbes Regional Hospital, Monroeville, Pennsylvania
  - Alle-Kiski Medical Center, Natrona Heights, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Clinic-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Susquehanna Cancer Center, Williamsport, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Kent County Hospital, Warwick, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville CCOP, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Cancer Centers of the Carolinas-Greer Medical Oncology, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Conklin Regional Cancer Center, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Blue Ridge Medical Specialists PC, Bristol, Tennessee
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Texas Cancer Center, Abilene, Texas
  - Texas Oncology PA - Amarillo, Amarillo, Texas
  - Texas Oncology-Arlington South, Arlington, Texas
  - Texas Oncology PA Beaumont, Beaumont, Texas
  - Texas Oncology PA - Bedford, Bedford, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Texas Cancer Center - Medical City Dallas, Dallas, Texas
  - Texas Health Presbyterian Hospital Dallas, Dallas, Texas
  - Texas Oncology Methodist Charlton Cancer Center, Dallas, Texas
  - Texas Oncology PA, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - Texas Oncology-El Paso, El Paso, Texas
  - Texas Oncology-Flower Mound, Flower Mound, Texas
  - Texas Oncology Fort Worth at 12th Avenue, Fort Worth, Texas
  - Texas Oncology - Garland, Garland, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Texas Oncology - Lewisville, Lewisville, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Texas Oncology-McAllen, McAllen, Texas
  - Texas Cancer Center - Mesquite, Mesquite, Texas
  - Texas Oncology-Midland Allison Cancer Center, Midland, Texas
  - Texas Oncology-Paris, Paris, Texas
  - North Texas Regional Cancer Center, Plano, Texas
  - Scott and White Healthcare Round Rock, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Cancer Care Centers of South Texas- Northeast, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - US Oncology Research LLC-The Woodlands, The Woodlands, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology PA, Waco, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Mountainview Medical, Berlin Corners, Vermont
  - University of Vermont, Burlington, Vermont
  - Rutland Regional Medical Center, Rutland, Vermont
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists-Fairfax, Fairfax, Virginia
  - Kaiser Permanente - Fair Oaks Medical Center, Fairfax, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Community Memorial Health Center, South Hill, Virginia
  - Peninsula Cancer Institute-Cancer Specialists of Tidewater, Virginia Beach, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - Shenandoah Oncology Associates PC, Winchester, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Auburn Regional Medical Center, Auburn, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison Bremerton Hematology and Oncology, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Puget Sound Cancer Center, Edmonds, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Cascade Cancer Center, Kirkland, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Harrison Poulsbo Hematology and Oncology, Poulsbo, Washington
  - Good Samaritan Community Hospital, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health, Seattle, Washington
  - Group Health Cooperative, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center, Spokane, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Allenmore Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - Saint Clare Hospital, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Northwest Cancer Specialists, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - City Hospital, Martinsburg, West Virginia
  - West Virginia University, Morgantown, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Wheeling Hospital, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Midelfort Clinic-Clairemont Campus, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital - Luther Campus, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital - ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Geyer CE Jr, Blum JL, Yothers G, Asmar L, Flynn PJ, Robert NJ, Hopkins JO, O'Shaughnessy JA, Rastogi P, Puhalla SL, Hilton CJ, Dang CT, Gomez HL, Vukelja SJ, Lyss AP, Paul D, Brufsky AM, Colangelo LH, Swain SM, Mamounas EP, Wolmark N. Long-Term Follow-Up of the Anthracyclines in Early Breast Cancer Trials (USOR 06-090, NSABP B-46-I/USOR 07132, and NSABP B-49 [NRG Oncology]). J Clin Oncol. 2024 Apr 20;42(12):1344-1349. doi: 10.1200/JCO.23.01428. Epub 2024 Feb 9. PMID 38335467